CLINICAL TRIAL: NCT06129591
Title: The Effects of Topical Cannabidiol on Paramedian Forehead Flap Scar Healing: A Split Scar Study (TOPSCAR)
Brief Title: Topical CBD Scar Healing Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OU-SCC-TOPSCAR
Record Dates: First submitted 2023-10-24; First posted 2023-11-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Paramedian Forehead Flap
Keywords: CBD oil; Paramedian Forehead Flap Reconstruction; silicone patch

STUDY DESIGN:
Intervention Model Description: This double arm, open label, single-site pilot trial aims to evaluate the feasibility of using topical CBD oil on paramedian forehead scars to determine if there is an improved outcome in the appearance of the scar.
Who Masked: Outcomes Assessor
Masking Description: The patient will know which part of the scar receives the silicone patch or silicone patch plus CBD because CBD requires separate oil application before the patch. However, the reviewing physicians will be blinded when assessing post-operative photos and using the SCAR scale.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Split-scar randomized trial arm with CBD oil (Experimental): The study targets the vertical forehead scar, treating half with CBD oil and a silicone patch (experimental).
  Interventions: Drug: Vantage Hemp CBD Isolate + Silicone patch
- Split-scar randomized trial arm without CBD oil (Placebo Comparator): The study targets the vertical forehead scar, treating the other scar half with a silicone patch (control).
  Interventions: Drug: Silicone patch

INTERVENTIONS:
Drug: Vantage Hemp CBD Isolate + Silicone patch — The study intervention is prospective in nature. This "split scar" study directly compares two parts of the healing scar during clinic visits. Photos will be taken at each visit to track progress. Assessments will be done over a period of around 7 months using the Modified Patient and Observer Scar Assessment Scale, followed by blinded photo evaluations using the Scar Cosmesis and Rating Scale.
  Arms: Split-scar randomized trial arm with CBD oil
Drug: Silicone patch — Standard of care silicone patch will be used as the control part of the split scar study. This "split scar" study directly compares two parts of the healing scar during clinic visits. Photos will be taken at each visit to track progress. Assessments will be done over a period of around 7 months using the Modified Patient and Observer Scar Assessment Scale, followed by blinded photo evaluations using the Scar Cosmesis and Rating Scale.
  Arms: Split-scar randomized trial arm without CBD oil

SUMMARY:
The purpose of this study is to find out what effects (good and bad) that cannabidiol (CBD) has on scar healing and appearance in patients who have undergone paramedian forehead flap reconstruction.

DETAILED DESCRIPTION:
The patient will be asked to apply a silicone patch to half of the scar and experimental ointment (CBD oil ointment) with silicone patch) to the other half of the scar on their forehead. They will be randomized to which half of the scar the ointment will be applied. Neither they nor their physician will choose which half of the scar will have the experimental ointment applied. Specific instructions will be given to the patient on how to apply each drug (the silicone patch to one segment of the scar and the CBD with silicone patch to the other segment of the scar). They will apply the treatments twice a day for 2 months and, at their follow-up appointments, complete two questionnaires about how the scar is healing. Photographs of the scars will be taken at each visit and will be evaluated to determine if there is an improved outcome in the appearance of the scar.

ELIGIBILITY:
Inclusion Criteria

* Patients that are adults (18+) of all genders and ethnicities who have undergone a PMFF (Paramedian forehead flap) will be considered for this study.
* English-speaking patients

Exclusion Criteria

* Patients younger than 18 years of age
* Non-English speaking patients
* Patients with known allergies to CBD
* Pregnant women
* Prisoners
* Patients with moderate to severe hepatic impairment
* A history of suicidal ideation and behavior within the last 6 months
* Patients with severe depression
* Who anticipate coadministration of other CNS depressants including alcohol that could potentiate the sedating effects of the drug
* Patients with a history of severe hypersensitivity reactions to adhesives
* Patients who anticipate coadministration of potentially hepatotoxic drugs
* Patients who anticipate coadministration of sensitive CYP2C19 substrates per labeling

Termination criteria

* There will be immediate termination from the study if any allergic response to the CBD/silicone combination occurs or if the topical application of CBD/silicone significantly worsens the scar outcome at the Follow Up 2 visit or at any subsequent visit.
* Subject will not receive any additional CBD doses if they experience an adverse event assessed as ≥ Grade 3 (including hepatotoxicities and hematologic adverse events, ≥ Grade 2 for the system-organ class of Cardiac Disorders) according to CTCAE v5. They will remain on study in follow-up until the adverse event resolves or stabilizes.
* If the patient voluntarily requests cessation in the study.
* Pregnancy
* Increase in serum transaminases (ALT/AST) to above three times the upper limit of normal or increase in total bilirubin to above two times the upper limit of normal.
* If a subject experiences worsening depression or suicidal ideation or behavior, the participant will be discontinued from treatment with CBD and immediately referred to a mental health professional. The decision to resume treatment with CBD will be made in collaboration with a mental health professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of subjective and objective effects of CBD on the outcomes of healing scars. | 2 years
  Proportion of patients who have a positive effect using CBD oil in combination with the silicone patch. This will be assessed using the Scar Cosmesis Assessment and Rating (SCAR) scale to determine the impact of CBD oil and silicon patch combo. This photographic evaluation of scare will be done over a period of around 7 months to evaluate the scar outcomes, using the scoring system with minimum score of 0 (being best possible outcome) and maximum score of 13 (worst possible scar outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mims, M.D., Ph.D., Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No